CLINICAL TRIAL: NCT03779672
Title: Randomized Double-blind Placebo-controlled Trial of Memantine Hydrochloride for the Treatment of Childhood-onset Epileptic Encephalopathies
Brief Title: Memantine for Epileptic Encephalopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kenneth Myers, MD (Other)
Responsible Party: Sponsor-Investigator, Kenneth Myers, MD, Assistant Professor (Clinical), Neurologist Pediatrician, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22838
Record Dates: First submitted 2018-12-05; First posted 2018-12-19 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Epileptic Encephalopathy, Childhood-Onset
Keywords: Memantine; N-methyl-D-aspartate receptor; Serum inflammatory; Seizure
MeSH Terms: conditions — Seizures | interventions — Memantine

STUDY DESIGN:
Intervention Model Description: Monocentric, Off-Label Use, Randomized, crossover, Double-blinded Placebo vs Memantine.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded Placebo vs Memantine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Memantine Hydrochloride 10 mg Placebo (Active Comparator): Blue colour capsules, for oral administration, containing 5 mg of active memantine or matching placebo for oral administration.
  Dose regimen:
  Memantine Hydrochloride
  * Week #1: 5 mg id (am), 1 caps
  * Week #2: 5 mg bid (am and pm), 2 caps
  * Weeks #3-6: 5 mg am & 2x 5 mg pm, 3 caps
  Washout (Weeks #7-8)
  Placebo
  * Week #9: id (am), 1 caps
  * Week #10: bid (am and pm), 2 caps
  * Weeks #11-14: 1 caps am & 2 caps pm, 3 caps
  Interventions: Drug: Memantine Hydrochloride 10 mg
- Placebo Memantine Hydrochloride 10 mg (Placebo Comparator): Placebo
  * Week #1: id (am), 1 caps
  * Week #2: bid (am and pm), 2 caps
  * Weeks #3-6: 1 caps am & 2 caps pm, 3 caps
  Washout (Weeks #7-8) Memantine Hydrochloride
  * Week #9: 5 mg id (am), 1 caps
  * Week #10: 5 mg bid (am and pm), 2 caps
  * Weeks #11-14: 5 mg am & 2x 5 mg pm, 3 caps
  Interventions: Drug: Memantine Hydrochloride 10 mg

INTERVENTIONS:
Drug: Memantine Hydrochloride 10 mg — * Week #1: 5 mg id (am), 1 caps
  * Week #2: 5 mg bid (am and pm), 2 caps
  * Weeks #3-6: 5 mg am & 2x 5 mg pm, 3 caps
  * Weeks #7-8: Washout
  Placebo
  * Week #9: id (am), 1 caps
  * Week #10: bid (am and pm), 2 caps
  * Weeks #11-14: 1 caps am & 2 caps pm, 3 caps
  OR Placebo
  * Week #1: id (am), 1 caps
  * Week #2: bid (am and pm), 2 caps
  * Weeks #3-6: 1 caps am & 2 caps pm, 3 caps
  * Weeks #7-8: Washout
  Memantine
  * Week #9: 5 mg id (am), 1 caps
  * Week #10: 5 mg bid (am and pm), 2 caps
  * Weeks #11-14: 5 mg am & 2x 5 mg pm, 3 caps
  Other Names: PrSANDOZ MEMANTINE FCT10 mg Drug Identification Number (DIN) 02375532

SUMMARY:
This study will evaluate the potential benefit of memantine hydrochloride as treatment for children with epileptic encephalopathy using a double-blind placebo-controlled cross-over design.

DETAILED DESCRIPTION:
Memantine, a drug approved for Alzheimer's dementia, exerts its therapeutic effect through its action as a low to moderate affinity non-competitive (open channel) N-methyl-D-aspartate receptor (NMDA-R) antagonist, which binds preferentially to the NMDA receptor-operated cation channels. It blocks the effects of persistently elevated levels of glutamate that may lead to neuronal dysfunction. Memantine may also have anti-inflammatory effects. Memantine has been used off-label in children and adolescents with autism spectrum disorder, to improve the cognitive impairment.

Epileptic encephalopathy, as well as other forms of epilepsy, may occur as a result of multiple etiologies, including genetic and inflammatory pathologies. Ion channels were long considered to be implicated in genetic epilepsy. Indeed one of the many possible causes of epilepsy is NMDA receptor dysfunction.

In the present study, the investigators plan to investigate the potential benefit of memantine as a treatment for epileptic encephalopathy. A double-blind placebo-controlled cross-over design will be used, with participants receiving 6 weeks of memantine and 6 weeks of placebo, with a 2-week washout period in between.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained
* Age 6-18 years (Weight ≥ 20 kg)
* Clinical diagnosis of epileptic encephalopathy

  * Subject with epilepsy and developmental impairment;
  * Epileptic activity itself contributes to severe cognitive and behavioural impairments
  * Patients will typically have already have trialed at least two standard therapies
* Females of childbearing age:
* Negative urinary pregnancy test at screening
* Agree to use effective contraception for the duration of the study

Exclusion Criteria:

* Inability of a parent or legal guardian to give informed consent for any reason.
* Known hypersensitivity to memantine hydrochloride
* Taking concomitant Amantadine, Ketamine or Dextromethorphan, Cimetidine, Ranitidine, Procainamide, Quinidine, Quinine, Hydrochlorothiazide, Anticholinergics, L-dopa, Anticoagulant,
* Any degree of renal impairment

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
Rate of Responder versus Non-Responder Status with Memantine | Week 6 or 14
  "Responder" defined as having ≥ 2 of (1) EEG improvement, (2) decreased seizure frequency, (3) cognitive improvement, (4) caregiver impression of improvement, (5) Serum Inflammatory Markers Change. These outcomes are individually defined in detail in the secondary outcomes below.
  Description of the primary variable(s) The primary efficacy endpoint is the composite cluster of the first occurrence, over the duration of study (randomization to study end date inclusive), of the EE improvement.
Rate of Responder versus Non-Responder Status with Placebo | Week 6 or 14
  "Responder" defined as having ≥ 2 of (1) EEG improvement, (2) decreased seizure frequency, (3) cognitive improvement, (4) caregiver impression of improvement, (5) Serum Inflammatory Markers Change. These outcomes are individually defined in detail in the secondary outcomes below.
  Description of the primary variable(s) The primary efficacy endpoint is the composite cluster of the first occurrence, over the duration of study (randomization to study end date inclusive), of the EE improvement.

SECONDARY OUTCOMES:
EEG Change with Memantine | Week 6 or 14
  EEG improvement EEG Change: EEG is not a quantitative measure, and there are many possible different patterns that may be seen in epileptic encephalopathy. In general, improvement usually involves (a) background activity changing to more closely resemble the expected background activity for the patient's age, and/or (b) decrease in frequency of epileptiform activity. The electroencephalographer will compare EEGs to the baseline study, and will score as (1) Interval worsening, (2) No significant change, or (3) Interval improvement.
  We will be assessing all the frequencies usually assessed on a routine EEG (delta, theta, alpha and beta). The frequency range assessed will be 1-70 Hz.
EEG Change with Placebo | Week 6 or 14
  EEG Change: EEG is not a quantitative measure, and there are many possible different patterns that may be seen in epileptic encephalopathy. In general, improvement usually involves (a) background activity changing to more closely resemble the expected background activity for the patient's age, and/or (b) decrease in frequency of epileptiform activity. The electroencephalographer will compare EEGs to the baseline study, and will score as (1) Interval worsening, (2) No significant change, or (3) Interval improvement.
  EEG improvement We will be assessing all the frequencies usually assessed on a routine EEG (delta, theta, alpha and beta). The frequency range assessed will be 1-70 Hz.
Seizure Frequency Change with Memantine | Week 6 or 14
  Reduction in seizure frequency Seizure Frequency Change: Participants will keep seizure diaries throughout the study. If the frequency of seizures decreases by > 50% from the baseline frequency, they will be classified as having a significant reduction in seizure frequency.
Seizure Frequency Change with Placebo | Week 6 or 14
  Reduction in seizure frequency Seizure Frequency Change: Participants will keep seizure diaries throughout the study. If the frequency of seizures decreases by > 50% from the baseline frequency, they will be classified as having a significant reduction in seizure frequency.
Cognitive Function Change with Memantine | Week 6 or 14
  Definite improvement in cognitive functioning by neuropsychological testing Cognitive Cognitive Function Change: Participants will see a neuropsychologist at baseline and at the conclusion of each treatment period. The precise testing used will be to the discretion of the neuropsychologist, based on the participant's cognitive capabilities. The neuropsychologist will compare to the baseline assessment and determine if there has been a significant change, based on her experience using these testing protocols in the given age range. The neuropsychologist will score as (1) Interval worsening, (2) No significant change, or (3) Interval improvement.
Cognitive Function Change with Placebo | Week 6 or 14
  Definite improvement in cognitive functioning by neuropsychological testing Cognitive Cognitive Function Change: Participants will see a neuropsychologist at baseline and at the conclusion of each treatment period. The precise testing used will be to the discretion of the neuropsychologist, based on the participant's cognitive capabilities. The neuropsychologist will compare to the baseline assessment and determine if there has been a significant change, based on her experience using these testing protocols in the given age range. The neuropsychologist will score as (1) Interval worsening, (2) No significant change, or (3) Interval improvement.
Caregiver Impression of Change with Memantine | Week 6 or 14
  Subjective perception of improvement by parents Caregiver Impression of Change: At the conclusion of each treatment period, caregivers will be asked the following question: "Compared to before the study, do you feel the overall functioning of your child (including seizure control, development and quality of life) is (1) Improved, (2) No Change, or (3) Worsened.
Caregiver Impression of Change with Placebo | Week 6 or 14
  Subjective perception of improvement by parents Caregiver Impression of Change: At the conclusion of each treatment period, caregivers will be asked the following question: "Compared to before the study, do you feel the overall functioning of your child (including seizure control, development and quality of life) is (1) Improved, (2) No Change, or (3) Worsened.
Serum Inflammatory Markers Change with Memantine | Week 6 or 14
  Changes in serum inflammation Serum inflammatory markers: C Reactive Protein (CRP), Erythrocyte Sedimentation Rate (ESR) and interleukin-6 (IL-6). CRP and ESR are commonly-used clinical measures of inflammation, and IL-6 was found to be elevated in some epileptic encephalopathies in one study (van den Munckhof et al., 2016). Levels will be compared following each treatment period, to the baseline value.
Serum Inflammatory Markers Change with Placebo | Week 6 or 14
  Changes in serum inflammation Serum inflammatory markers: C Reactive Protein (CRP), Erythrocyte Sedimentation Rate (ESR) and interleukin-6 (IL-6). CRP and ESR are commonly-used clinical measures of inflammation, and IL-6 was found to be elevated in some epileptic encephalopathies in one study (van den Munckhof et al., 2016). Levels will be compared following each treatment period, to the baseline value.

OTHER OUTCOMES:
Adverse events | Week 16
  Participants will be asked at all visits to report any possible adverse events, including those requiring emergent treatment. Adverse events will be classified as "clinically significant" or "not clinically significant" with respect to the likelihood that they are related to use of the investigational drug. The frequency of adverse events will be determined during the period receiving memantine and the period receiving placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- Children Hospital - MUHC, Montreal, Quebec, Canada

REFERENCES:
- [Background] van den Munckhof B, de Vries EE, Braun KP, Boss HM, Willemsen MA, van Royen-Kerkhof A, de Jager W, Jansen FE. Serum inflammatory mediators correlate with disease activity in electrical status epilepticus in sleep (ESES) syndrome. Epilepsia. 2016 Feb;57(2):e45-50. doi: 10.1111/epi.13274. Epub 2015 Dec 14. PMID 26666401
- [Derived] Schiller K, Berrahmoune S, Dassi C, Corriveau I, Ayash TA, Osterman B, Poulin C, Shevell MI, Simard-Tremblay E, Sebire G, Myers KA. Randomized placebo-controlled crossover trial of memantine in children with epileptic encephalopathy. Brain. 2023 Mar 1;146(3):873-879. doi: 10.1093/brain/awac380. PMID 36256600